CLINICAL TRIAL: NCT02896569
Title: Clinical Evaluation of the Tolerability of Using a Post Treatment Topical Adjuvant Combination Following Fractional Radiofrequency Ablation Using the Venus Viva
Brief Title: Tolerability of Using a Post-Treatment Topical Adjuvant Combination Following Fractional Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS0116
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Skin Disorders
Keywords: resurfacing; ablation
MeSH Terms: conditions — Skin Diseases | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical combination therapy (Experimental): Application of human bone marrow stem cell derived growth factor and cytokines serum followed by a botanical lipid-based occlusive immediately post-radio-frequency treatment of the face
  Interventions: Other: Topical combination therapy
- Standard of care (No Intervention): No topical therapies for 24 hours post-radio-frequency treatment of the face

INTERVENTIONS:
Other: Topical combination therapy
  Other Names: SCR Complex; Bio Cel
  Arms: Topical combination therapy

SUMMARY:
The purpose of this study is to compare the tolerability of the application of a combination of a serum containing human bone marrow stem cell derived growth factor (SCR Complex) and cytokines and a botanical lipid-based occlusive (Bio Cel) immediately following fractional radiofrequency treatment using the Venus Viva versus standard of care.

DETAILED DESCRIPTION:
Randomized, open-label, multi-centre study to evaluate the tolerability of the application of a combination of a serum containing human bone marrow stem cell derived growth factor and cytokines (SCR Complex™) and a botanical lipid based occlusive (Bio Cel™) following facial fractional RF treatments using the Venus Viva™ SR system. Each subject will receive 2 treatments separated by a 3-week interval. Subjects will complete a VAS and Tolerability Scale immediately following each treatment. Telephone follow-up calls by the site will ask the subject to respond to the Self-Report Adverse Event Questionnaire 24 and 72 hours after the first treatment and 24 hours after the second treatment. Subjects will complete a Home Tolerability Scale 24 and 72 hours after the first treatment and 24 hours after the second treatment. Subjects will return for the final FU visit and be asked to respond to the Self-Report Adverse Event Questionnaire and complete the Home Tolerability Scale for 72 hours. The investigator will also evaluate the subject's improvement using the GAIS at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a dermatological procedure requiring ablation and resurfacing of the facial skin utilizing the Venus Viva™ SR system.
* Women of child-bearing age are required to be using a reliable method of birth control prior to enrollment and throughout their participation in the study.
* Able to tolerate the treatment as determined by a test spot application(s).

Exclusion Criteria:

* Superficial metal or other implants in the treatment area
* Tattoos, permanent makeup, scars or piercings in the treatment area.
* Any active condition in the treatment area, such as sores, psoriasis, eczema and rash.
* Any surgical procedure in the treatment area within the last three months or before complete healing.
* Receiving therapies or medication that may interfere with the study treatment.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Reiz, BSc, Study Director — Venus Concept Ltd.
Locations (1):
- Dr. George Taylor, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Combination Therapy: Application of human bone marrow stem cell derived growth factor and cytokines serum followed by a botanical lipid-based occlusive immediately post-radio-frequency treatment of the face
  Topical combination therapy
Period: Overall Study
Arm/Group | Topical Combination Therapy | Standard of Care
Started | 25 | 24
Completed | 21 | 19
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Combination Therapy | Standard of Care | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants] — The protocol was amended to include subjects >/= 75 years of age.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 22 | 23 | 45
    >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 23 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 16 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Tolerability of Initial Treatment [Count of Participants; unit: Participants] — The primary endpoint of the study is the tolerability of the combination treatment vs standard of care treatment. This baseline measure of tolerability to the first treatment is the measure from which succeeding treatments were compared to . Population: Not all subjects had the initial treatment tolerability reported. Twenty-three subjects in each of the treatment groups reported the initial tolerability.
  Participants
    number analyzed (Participants) | 23 | 23 | 46
    Initial treatment - Very Tolerable | 11 | 7 | 18
    Initial Treatment - Tolerable | 11 | 16 | 27
    Initial Treatment - Having no opinion | 1 | 0 | 1
    Initial treatment - Intolerable | 0 | 0 | 0
    Initial treatment - Very intolerable | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject Treatment Tolerability Score Post Treatment 1 at 24hrs Post Treatment
Description: Tolerability 5-point Likert scale where 4 - Very Tolerable, 3 - Tolerable, 2 - Having no opinion, 1 - Intolerable and 0 - very intolerable; The higher the score, the more tolerable the subject indicates the treatment is.
Time Frame: 24hr post treatment one
Population: Not all subjects only responded to telephone request for tolerability at 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 22 | 21
Participants
  Tx 1 at 24 hr Very Tolerable | 15 | 18
  Tx 1 at 24 hr Tolerable | 7 | 3
  Tx 1 at 24 hr Having No Opinion | 0 | 0
  Tx 1 at 24 hr InTolerable | 0 | 0
  Tx 1 at 24 hr Very Intolerable | 0 | 0

2. Primary Outcome: Subject Treatment Tolerability Score Post Treatment 1 at 72hrs Post Treatment
Description: as for outcome 1
Time Frame: 72 hrs post treatment one
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 20 | 18
Participants
  Tx 1 at 72 hr - Very Tolerable | 17 | 17
  Tx 1 at 72 hr - Tolerable | 3 | 0
  Tx 1 at 72 hr Having No Opinion | 0 | 0
  Tx 1 at 72 hr InTolerable | 0 | 1
  Tx 1 at 72 hr Very Intolerable | 0 | 0

3. Primary Outcome: Subject Treatment Tolerability Score Post Treatment 2 at 24hrs Post Treatment
Description: as for outcome 1
Time Frame: 24hr post treatment two
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 21 | 18
Participants
  Tx 2 at 24 hr - Very Tolerable | 18 | 14
  Tx 2 at 24 hr - Tolerable | 3 | 4
  Tx 2 at 24 hr Having No Opinion | 0 | 0
  Tx 2 at 24 hr InTolerable | 0 | 0
  Tx 2 at 24 hr Very Intolerable | 0 | 0

4. Primary Outcome: Subject Treatment Tolerability Score Post Treatment 2 at 72 Hrs Post Treatment
Description: as for outcome 1
Time Frame: 72hr post treatment two
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 21 | 18
Participants
  Tx 2 at 72 hr - Very Tolerable | 19 | 17
  Tx 2 at 72 hr - Tolerable | 2 | 1
  Tx 2 at 72 hr Having No Opinion | 0 | 0
  Tx 2 at 72 hr InTolerable | 0 | 0
  Tx 2 at 72 hr Very Intolerable | 0 | 0

5. Secondary Outcome: Visual Analog Scale
Description: 10 cm Subject discomfort scale where 10 cm indicates 'Pain as bad as it can be' and 0 cm indicates there is no pain at all associated with the application of the treatment. Zero pain means a better outcome. Subjects were categorized as to having no pain (0 - 0.4cm), mild pain (0.5 - 4.4cm), moderate pain (4.5 - 7.4cm) and severe pain (7.5 - 10cm).
Time Frame: immediately following radio-frequency treatment
Population: Not all subjects reported VAS for each treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 25 | 23
Participants
  Treatment 1: No pain (0 - 0.4cm) | 1 | 1
  Treatment 1: Mild Pain (0.5 - 4.4 cm) | 16 | 13
  Treatment 1: Moderate Pain (4.5 - 7.4 cm) | 6 | 7
  Treatment 1: Severe Pain (7.5 - 10 cm) | 2 | 2
  Treatment 2: number analyzed (Participants) | 21 | 19
  Treatment 2: No pain (0 - 0.4cm) | 2 | 0
  Treatment 2: Mild Pain (0.5 - 4.4 cm) | 11 | 9
  Treatment 2: Moderate Pain (4.5 - 7.4 cm) | 7 | 8
  Treatment 2: Severe Pain (7.5 - 10 cm) | 1 | 2

6. Secondary Outcome: Fitzpatrick Wrinkle and Elastosis Scale
Description: Investigator assessment of improvement in wrinkles and elastosis where Class I indicates fine wrinkles, Class II indicates fine to moderate depth wrinkles with a moderate number of lines and Class III indicates fine to deep wrinkles, numerous lines with or without redundant skin folds with a score of 1 - 3 (Mild) indicates fine texture changes with subtly accentuated skin lines, a score of 4 - 6 (Moderate) indicates distinct papular elastosis ([indvidual papules with yellow translucency under direct lighting] and dyschromia and a score of 7 - 9 (Severe) indicates multipapular and confluent elastosis [thickened yellow and pallid] approaching or consistent with cutis rhomboidalis. A lower class and a lower score means a better outcome. Subjects were divided into 3 categories - No change in FWES score, change in FWES score by one and non-evaluable.
Time Frame: change in appearance of wrinkles from baseline and at end of study, average of 24 days
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 25 | 24
Participants
  No change in FWES score | 23 | 23
  FWES score increased by one | 2 | 0
  Non-evaluable | 0 | 1

7. Secondary Outcome: Global Aesthetic Improvement Scale
Description: Investigator assessment of aesthetic improvement where 1 shows exceptional improvement, 2 shows very improved, 3 shows improvement, 4 shows unchanged and 5 indicates that the subject appearance has worsened. A low score means a better outome. Subjects were categorized to either GAIS improved or GAIS no change.
Time Frame: change in skin appearance between baseline and at end of study, average of 24 days
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Combination Therapy | Standard of Care
Number analyzed (Participants) | 20 | 23
Participants
  GAIS Improved | 12 | 14
  GAIS No Change | 8 | 9

ADVERSE EVENTS:
Time Frame: The study collected adverse event data for 3 months 4 days.
Arm/Group | Topical Combination Therapy | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02896569/Prot_SAP_000.pdf